CLINICAL TRIAL: NCT02384382
Title: A PHASE 2, OPEN-LABEL, SINGLE-ARM STUDY OF 18F-SODIUM FLUORIDE PET/CT BONE IMAGING IN ENZALUTAMIDE-TREATED CHEMOTHERAPY-NAÏVE PATIENTS WITH BONE-METASTATIC CASTRATION-RESISTANT PROSTATE CANCER
Brief Title: A Positron Emission Tomography/Computed Tomography (PET/CT) Bone Imaging Study in Patients Receiving Enzalutamide for Castration-Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDV3100-18; C3431012 (Other: Alias Study Number)
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Prostate Carcinoma Metastatic to the Bone; Castration Resistant Prostate Cancer
Keywords: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide monotherapy (Experimental): Enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: MDV3100; Xtandi

SUMMARY:
The purpose of this study is to evaluate 18F-sodium fluoride positron-emission tomography / computed tomography (18F-NaF PET/CT) imaging as a method for determining treatment response in metastatic bone lesions in patients who are receiving enzalutamide for castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, or signet cell or small cell features;
* Presence of bone metastatic disease as assessed by at least two lesions on whole body metastable technetium-methylene diphosphonate (99mTc-MDP) bone scintigraphy;
* Throughout the study, ongoing androgen deprivation therapy with a luteinizing hormone-releasing hormone (LHRH) analogue or prior bilateral orchiectomy (medical or surgical castration);
* Testosterone ≤ 1.73 nmol/L (≤ 50 ng/dL) at screening;
* Progressive disease on androgen deprivation therapy at screening defined as a minimum of two sequentially rising prostate-specific antigen (PSA) values (PSA1 < PSA2 < PSA3);
* The screening PSA (PSA3) must be ≥ 2 μg/L (≥ 2 ng/mL).

Exclusion Criteria:

* Prior enzalutamide, abiraterone acetate, aminoglutethimide, ketoconazole, radium Ra 223 dichloride or other bone-targeting radionuclides, or cytotoxic chemotherapy in the CRPC setting for the treatment of prostate cancer or participation in a clinical trial of an investigational agent that inhibits the androgen receptor or androgen synthesis (unless treatment was placebo);
* Treatment with hormonal therapy (eg, androgen receptor inhibitors, 5-alpha reductase inhibitors) or biologic therapy for prostate cancer (other than LHRH analogue therapy) within 4 weeks before enrollment;
* Initiation of new treatment with denosumab, bisphosphonates, or systemic corticosteroids for treatment of prostate cancer within 4 weeks before enrollment;
* Use of an investigational agent within 4 weeks before the screening visit;
* Radiation therapy to bone within 4 weeks before enrollment;
* Use of opiate analgesics for prostate cancer pain within 4 weeks before enrollment;
* Screening 99mTc-MDP bone scintigraphy showing a superscan;
* Visceral (eg, lung, liver) metastatic disease. Adenopathy is allowed;
* Current or previously treated brain metastasis or active leptomeningeal disease;
* History of seizure any time in the past for any reason or any condition that may predispose to seizures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Wimr Pet/Ct, Madison, Wisconsin
  - UW Clinical Sciences Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kyriakopoulos CE, Heath EI, Ferrari A, Sperger JM, Singh A, Perlman SB, Roth AR, Perk TG, Modelska K, Porcari A, Duggan W, Lang JM, Jeraj R, Liu G. Exploring Spatial-Temporal Changes in 18F-Sodium Fluoride PET/CT and Circulating Tumor Cells in Metastatic Castration-Resistant Prostate Cancer Treated With Enzalutamide. J Clin Oncol. 2020 Nov 1;38(31):3662-3671. doi: 10.1200/JCO.20.00348. Epub 2020 Sep 8. PMID 32897830

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide 160 Milligram (mg) (18F-NaF PET/CT): Chemotherapy naive participants with progressive bone-metastatic castration-resistant prostate cancer (CRPC) were enrolled to receive enzalutamide 160 milligram (mg) per day as 4 capsules (each capsule of 40 mg), orally, once daily. 18F-sodium fluoride positron-emission tomography/computed tomography bone imaging (18F-NaF PET/CT) was evaluated to determine treatment response in metastatic bone lesions of enrolled participants in the study. Maximum treatment exposure was 34.1 months.
Period: Overall Study
Arm/Group | Enzalutamide 160 Milligram (mg) (18F-NaF PET/CT)
Started | 23
Completed | 0
Not Completed | 23
Not completed — Transitioned to study-NCT02960022 | 5
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Disease progression | 16

BASELINE CHARACTERISTICS:
Population: As treated population included all enrolled participants who received any amount of study medication.
Groups:
- Enzalutamide 160 mg (18F-NaF PET/CT): Chemotherapy naive participants with progressive bone-metastatic CRPC were enrolled to receive enzalutamide 160 mg per day as 4 capsules (each capsule of 40 mg), orally, once daily. 18F-NaF PET/CT was evaluated to determine treatment response in metastatic bone lesions of enrolled participants in the study. Maximum treatment exposure was 34.1 months.
Arm/Group | Enzalutamide 160 mg (18F-NaF PET/CT)
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least (>=) 1 Responding Bone Lesion Assessed by Total Sodium Fluoride (NaF) Standardized Uptake Value [SUVtotal] at Third 18F-NaF PET/CT Imaging (NaF-3) Schedule
Description: Bone lesion responded: if its change from baseline in SUVtotal is below limit of agreement (LOA, no specific value, based upon test/retest analysis using software). SUVtotal: total NaF uptake,indicated tumor burden across all bone lesions/in individual lesions reflecting bone-metastatic prostate cancer.NaF-3 performed on any of these: 1) prostate-specific antigen (PSA) progression(increase of >=25% and absolute increase of >=2.0 ng/mL above nadir); 2) bone progressive disease(PD)(appearance of >=2 new lesions after screening assessed by technetium Tc 99m medronate [99mTc-MDP] bone scintigraphy); 3) soft tissue PD; 4) clinically relevant progression by investigator; 5) at 2 years without progression after treatment initiation. PD, RECIST1.1:>=20% increase in sum of diameters of target lesions,(reference smallest sum on study, included baseline sum if that is smallest on study),relative increase of 20%,sum of diameters indicated absolute increase of >=5mm, appearance of >=1 new lesions.
Time Frame: At NaF-3 schedule: at time of PSA, or radiographic(bone or soft tissue), or clinically relevant progression, or at 2years without progression after treatment initiation, whichever occurred first(From first dose of study drug up to maximum of 34.1 months)
Population: Analysis population included all enrolled participants who received any amount of study medication and who also have non-missing scans at both NaF-1 and NaF-3. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide 160 mg (18F-NaF PET/CT)
Number analyzed (Participants) | 22
percentage of participants | 100.0 [84.6 to 100.0]

2. Secondary Outcome: Mean Heterogeneity of Response Across All Bone Lesions as Measured by Global Heterogeneity of NaF Standardized Uptake (SUVhetero) Score at Third 18F-NaF PET/CT Imaging (NaF-3) Schedule
Description: Global SUVhetero score:Sum of(SUVmean of each lesion minus global SUVmean of all lesion)^2/number of lesions,measure of heterogeneity of tumor activity across all bone lesions.SUVmean(mean NaF uptake)indicated average activity of each lesions.Real limits for SUVhetero score ranged:0(minimum) to infinite(maximum).Higher global SUVhetero score:more heterogeneity in bone lesion activity.NaF-3 performed on any of these 1)PSA progression(increase of>=25% and absolute increase of>=2.0ng/mL above nadir);2)bone PD(appearance of>=2 new lesions after screening assessed by 99mTc-MDP bone scintigraphy);3)soft tissue PD(RECIST1.1);4)clinically relevant progression by investigator;5)at 2years without progression after treatment initiation.PD perRECIST1.1:>=20%increase in sum of diameters of target lesions,(reference smallest sum on study,this included baseline sum if that is smallest on study),relative increase of20%,sum of diameters indicated absolute increase of>=5mm,appearance of>=1 new lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: unit on SUVhetero score
Arm/Group | Enzalutamide 160 mg (18F-NaF PET/CT)
Number analyzed (Participants) | 22
unit on SUVhetero score | 3.9 (3.17)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study treatment or initiation of cytotoxic chemotherapy, (lutamide- bicalutamide, nilutamide,or flutamide), or initiation of new investigational therapy, whichever occurred first (up to 35.1 months)
Description: Same event may appear as adverse events (AEs) and serious adverse events (SAEs), what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non serious event during study. As treated population included all enrolled participants who received any amount of study medication.
Groups:
- Enzalutamide 160 mg: Chemotherapy naive participants with progressive bone-metastatic CRPC were enrolled to receive enzalutamide 160 mg per day as 4 capsules (each capsule of 40 mg), orally, once daily. 18F-NaF PET/CT was evaluated to determine treatment response in metastatic bone lesions of enrolled participants in the study. Maximum treatment exposure was 34.1 months.
Arm/Group | Enzalutamide 160 mg
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide 160 mg (N=23)
Mitral valve incompetence (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Completed suicide (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide 160 mg (N=23)
Anaemia (Blood and lymphatic system disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 2
Retinal haemorrhage (Eye disorders) | 1
Asthenia (General disorders) | 3
Chest pain (General disorders) | 3
Fatigue (General disorders) | 19
Gait disturbance (General disorders) | 1
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 2
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Procedural pain (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Parosmia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Stress urinary incontinence (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Cyst drainage (Surgical and medical procedures) | 1
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02384382/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT02384382/SAP_001.pdf